CLINICAL TRIAL: NCT05925517
Title: The Effect of Graded Motor Imagery on Pain and Function in Individuals With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The Effect of Graded Motor Imagery on Pain and Function in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Graded Motor Imagery
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis; Limitation, Mobility
Keywords: Pain; Knee Joint; Exercise; Range of Motion; Muscle Strength
MeSH Terms: conditions — Osteoarthritis, Knee; Mobility Limitation; Pain; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: In this prospective study, two treatment groups were formed to receive GMI and TENS.
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Motor Imagery (Experimental): Each patient in the Graded Motor Imagery group will receive a treatment protocol consisting of Graded Motor Imagery, conventional physiotherapy, and home exercises.
  Interventions: Other: Graded Motor Imagery (GMI); Other: Conventional Physiotherapy Program; Other: Home Exercise Protocol
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Each patient in the Transcutaneous Electrical Nerve Stimulation group will receive a treatment protocol consisting of Transcutaneous Electrical Nerve Stimulation, conventional physiotherapy, and home exercises.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Conventional Physiotherapy Program; Other: Home Exercise Protocol

INTERVENTIONS:
Other: Graded Motor Imagery (GMI) — GMI includes three stages. Each session will be 30 minutes, and the GMI program will span over 8 weeks. The first 3 weeks will focus on lateralization, followed by 3 weeks of motor imagery, and the final 2 weeks will involve mirror therapy.
  Lateralization: Patients will be asked to differentiate whether the extremities shown in the Recognise™ Knee application belong to the right or left side of their body.
  Motor Imagery: Patients will be instructed to imagine slowly and smoothly moving their affected extremities to the posture depicted in the photos in the Recognise™ Knee application and then returning to the starting position.
  Mirror Therapy: Using a mirror measuring 90x60 cm² placed between the lower extremities, patients will be instructed to progressively move only their unaffected extremity, then their affected extremity, and finally both extremities.
  Other Names: GMI
  Arms: Graded Motor Imagery
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — Application will be performed using a TENS device and four separate 2 × 2 inch self-adhesive electrodes. The current will be applied to the most painful area of the affected knee. The four self-adhesive electrodes will be positioned in a square pattern, approximately 5 cm apart, centered over the pain point. Conventional TENS will be applied for 30 minutes at a frequency of 100 Hz, pulse width of 100 μs, and intensity below 10% of the motor threshold.
  Other Names: TENS
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)
Other: Conventional Physiotherapy Program — The routine 60-minute program for OA patients in conventional physiotherapy includes warming up, core stability, pelvic and hip stability, gluteus medius strengthening, knee control and stability (knee flexion and extension control, lunge exercises), knee strengthening exercises (wall-assisted leg press with a ball, step-ups with elastic bands), and functional exercises.
Other: Home Exercise Protocol — The home exercises will include a warm-up consisting of a 10-minute walk at a normal pace on a flat surface while gently stretching the hamstring and calf muscles. The exercises will also involve straight leg raises, terminal knee extension, isometric contractions of the quadriceps femoris and adductor muscles using a pillow for support, toe raises, single-leg standing, toe taps, and quadriceps strengthening exercises included in the session.

SUMMARY:
The aim of this study is to investigate whether Graded Motor Imagery (GMI) application is as effective as Transcutaneous Electrical Nerve Stimulation (TENS) in individuals with knee osteoarthritis (OA). The objectives are to improve range of motion (ROM) and muscle strength, reduce pain and stiffness, increase pain pressure threshold, and enhance function and physical performance through GMI application.

DETAILED DESCRIPTION:
46 voluntary patients with knee OA, aged between 45-64 years will be randomly divided into two groups: GMI group and TENS group. Interventions will be applied for 8 weeks, 3 times a week (24 sessions). Both groups will receive conventional physiotherapy and home exercises in addition to GMI or TENS treatment. The patients will be assessed before, after treatment and six-week follow-up. Knee pain will be evaluated using the Visual Analog Scale (VAS), pressure pain threshold will be measured using an algometer, pain, function, and stiffness will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), active knee range of motion will be measured using a digital goniometer, muscle strength will be evaluated using a hand-held dynamometer, and function will be assessed using the Timed Up and Go Test.

ELIGIBILITY:
Inclusion Criteria:

* Minimum score of 24 on the Mini Mental State Examination (indicating no mild or severe dementia)
* Diagnosis of moderate unilateral knee osteoarthritis persisting for more than 12 months according to American College of Rheumatology (ACR) criteria
* Experience of pain with a severity rating of 3 or higher on the Visual Analog Scale (VAS) for activities such as stair climbing, sitting, and squatting, lasting for at least 6 months (moderate to severe pain)
* Age between 45 and 64 years
* Residing in the city where the study is conducted
* Ability to walk independently
* Presence of limitations in knee range of motion (ROM)
* Symptomatic and radiographically confirmed OA diagnosis of Kellgren and Lawrence grade I-III

Exclusion Criteria:

* Patients who are unwilling to participate in the study
* Patients presenting with secondary OA due to conditions such as rheumatoid arthritis, gout, septic arthritis, tuberculosis, tumor, trauma, hemophilia, major medical or psychiatric disorders, recent fractures, presence of effusion or open reduction and internal fixation in the knee
* Presence of a neuromuscular disease
* History of intra-articular injections in the past 6 months
* Patients undergoing medication changes
* Presence of any chronic illness that would hinder participation in the treatment program
* Participation in a physiotherapy program for OA in the last 12 weeks
* Movement limitations or limb deficiency in the contralateral lower extremity
* Presence of visual or hearing problems that would affect treatment adherence.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline
  Visual Analogue Scale (VAS) will be used to evaluate the severity of pain felt around the knee joint. Participants will be asked to mark the severity of the pain they feel (rest, activity and night) on a 10 cm horizontal line, from 0 (no pain) to 10 (unbearable pain).
Pain Intensity | After the 8-week intervention
  Visual Analogue Scale (VAS) will be used to evaluate the severity of pain felt around the knee joint. Participants will be asked to mark the severity of the pain they feel (rest, activity and night) on a 10 cm horizontal line, from 0 (no pain) to 10 (unbearable pain).
Pain Intensity | 6-week follow-up
  Visual Analogue Scale (VAS) will be used to evaluate the severity of pain felt around the knee joint. Participants will be asked to mark the severity of the pain they feel (rest, activity and night) on a 10 cm horizontal line, from 0 (no pain) to 10 (unbearable pain).
Pain Pressure Threshold | Baseline
  The pain pressure threshold will be measured using a algometer. The pain pressure threshold will be evaluated at two points while the patient is lying in a lateral position: 1. point located 2 cm below the medial edge of the patella, and 2. point located 2 cm below the lateral edge of the patella. The evaluator will position the algometer perpendicular to each point and apply gradual pressure at a constant rate of approximately 0.5 kg/cm2/s. The pressure will be increased until the participant reports feeling pain. Each point considered for analysis will be assessed three times, and the average value will be recorded.
Pain Pressure Threshold | After the 8-week intervention
  The pain pressure threshold will be measured using a algometer. The pain pressure threshold will be evaluated at two points while the patient is lying in a lateral position: 1. point located 2 cm below the medial edge of the patella, and 2. point located 2 cm below the lateral edge of the patella. The evaluator will position the algometer perpendicular to each point and apply gradual pressure at a constant rate of approximately 0.5 kg/cm2/s. The pressure will be increased until the participant reports feeling pain. Each point considered for analysis will be assessed three times, and the average value will be recorded.
Pain Pressure Threshold | 6-week follow-up
  The pain pressure threshold will be measured using a algometer. The pain pressure threshold will be evaluated at two points while the patient is lying in a lateral position: 1. point located 2 cm below the medial edge of the patella, and 2. point located 2 cm below the lateral edge of the patella. The evaluator will position the algometer perpendicular to each point and apply gradual pressure at a constant rate of approximately 0.5 kg/cm2/s. The pressure will be increased until the participant reports feeling pain. Each point considered for analysis will be assessed three times, and the average value will be recorded.
WOMAC Pain Subscale | Baseline
  The subscale can take a score between 0-20 and evaluates pain during walking on flat ground, going up and down stairs, standing, sitting and lying down.
WOMAC Pain Subscale | After the 8-week intervention
  The subscale can take a score between 0-20 and evaluates pain during walking on flat ground, going up and down stairs, standing, sitting and lying down.
WOMAC Pain Subscale | 6-week follow-up
  The subscale can take a score between 0-20 and evaluates pain during walking on flat ground, going up and down stairs, standing, sitting and lying down.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Baseline
  The WOMAC index will be used to evaluate pain, stiffness, and function. It contains 24 items scored from 0 to 4: 0=absent, 1=mild, 2=moderate, 3=severe, and 4=extreme.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | After the 8-week intervention
  The WOMAC index will be used to evaluate pain, stiffness, and function. It contains 24 items scored from 0 to 4: 0=absent, 1=mild, 2=moderate, 3=severe, and 4=extreme.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | 6-week follow-up
  The WOMAC index will be used to evaluate pain, stiffness, and function. It contains 24 items scored from 0 to 4: 0=absent, 1=mild, 2=moderate, 3=severe, and 4=extreme.
Range of Motion (ROM) | Baseline
  Knee ROM will be evaluated with a digital goniometer while the participants lie comfortably in the prone position while active knee joint motion will be evaluated. Evaluation will be performed with the pivot point following the lateral condyle of the femur, the fixed arm following the lateral midline of the femur, and the mobile arm following the fibula. The measurements will be repeated three times for the affected and unaffected side, and the best value between the measurements will be recorded.
Range of Motion (ROM) | After the 8-week intervention
  Knee ROM will be evaluated with a digital goniometer while the participants lie comfortably in the prone position while active knee joint motion will be evaluated. Evaluation will be performed with the pivot point following the lateral condyle of the femur, the fixed arm following the lateral midline of the femur, and the mobile arm following the fibula. The measurements will be repeated three times for the affected and unaffected side, and the best value between the measurements will be recorded.
Range of Motion (ROM) | 6-week follow-up
  Knee ROM will be evaluated with a digital goniometer while the participants lie comfortably in the prone position while active knee joint motion will be evaluated. Evaluation will be performed with the pivot point following the lateral condyle of the femur, the fixed arm following the lateral midline of the femur, and the mobile arm following the fibula. The measurements will be repeated three times for the affected and unaffected side, and the best value between the measurements will be recorded.
Isometric Muscle Strength | Baseline
  Flexion and extension isometric muscle strength of the knee will be assessed using a hand-held dynamometer. During the assessment, maximum voluntary contraction will be requested. Measurements will be repeated three times (5 seconds of contraction followed by 30 seconds of rest) for both affected and unaffected knees, and the average value will be recorded in Newtons (N). Patients will sit with their backs straight, arms crossed, hips flexed at 90°, and knees flexed at 30°, with their feet hanging off the side of the bed. The dynamometer will be placed on the anterior surface of the tibia, two fingers above the lateral malleolus.
Isometric Muscle Strength | After the 8-week intervention
  Flexion and extension isometric muscle strength of the knee will be assessed using a hand-held dynamometer. During the assessment, maximum voluntary contraction will be requested. Measurements will be repeated three times (5 seconds of contraction followed by 30 seconds of rest) for both affected and unaffected knees, and the average value will be recorded in Newtons (N). Patients will sit with their backs straight, arms crossed, hips flexed at 90°, and knees flexed at 30°, with their feet hanging off the side of the bed. The dynamometer will be placed on the anterior surface of the tibia, two fingers above the lateral malleolus.
Isometric Muscle Strength | 6-week follow-up
  Flexion and extension isometric muscle strength of the knee will be assessed using a hand-held dynamometer. During the assessment, maximum voluntary contraction will be requested. Measurements will be repeated three times (5 seconds of contraction followed by 30 seconds of rest) for both affected and unaffected knees, and the average value will be recorded in Newtons (N). Patients will sit with their backs straight, arms crossed, hips flexed at 90°, and knees flexed at 30°, with their feet hanging off the side of the bed. The dynamometer will be placed on the anterior surface of the tibia, two fingers above the lateral malleolus.
Mini Mental State Examination | Baseline
  The Mini-Mental State Examination (MMSE) will be used to assess the cognitive status of patients. It consists of 11 questions and is evaluated on a scale of 30 points. A score between 24-30 is considered normal, 18-23 indicates mild cognitive impairment, and a score of 17 or below is indicative of severe dementia. The MMSE assesses orientation, memory, attention, calculation, recall, language, motor function, perception, and visuospatial abilities.
Mini Mental State Examination | After the 8-week intervention
  The Mini-Mental State Examination (MMSE) will be used to assess the cognitive status of patients. It consists of 11 questions and is evaluated on a scale of 30 points. A score between 24-30 is considered normal, 18-23 indicates mild cognitive impairment, and a score of 17 or below is indicative of severe dementia. The MMSE assesses orientation, memory, attention, calculation, recall, language, motor function, perception, and visuospatial abilities.
Mini Mental State Examination | 6-week follow-up
  The Mini-Mental State Examination (MMSE) will be used to assess the cognitive status of patients. It consists of 11 questions and is evaluated on a scale of 30 points. A score between 24-30 is considered normal, 18-23 indicates mild cognitive impairment, and a score of 17 or below is indicative of severe dementia. The MMSE assesses orientation, memory, attention, calculation, recall, language, motor function, perception, and visuospatial abilities.
Timed Get Up and Go Test (TUG) | Baseline
  The test will be initiated with each participant sitting on a chair with their back supported, arms resting on their lap, and both feet flat on the floor. Participants will be timed using a stopwatch as they rise from the chair (45 cm in height), walk 3 meters as quickly and safely as possible, turn around, return to the chair, and sit down. The time taken for each participant to complete these tasks will be recorded using a stopwatch.
Timed Get Up and Go Test (TUG) | After the 8-week intervention
  The test will be initiated with each participant sitting on a chair with their back supported, arms resting on their lap, and both feet flat on the floor. Participants will be timed using a stopwatch as they rise from the chair (45 cm in height), walk 3 meters as quickly and safely as possible, turn around, return to the chair, and sit down. The time taken for each participant to complete these tasks will be recorded using a stopwatch.
Timed Get Up and Go Test (TUG) | 6-week follow-up
  The test will be initiated with each participant sitting on a chair with their back supported, arms resting on their lap, and both feet flat on the floor. Participants will be timed using a stopwatch as they rise from the chair (45 cm in height), walk 3 meters as quickly and safely as possible, turn around, return to the chair, and sit down. The time taken for each participant to complete these tasks will be recorded using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, PhD, Principal Investigator — Artvin Coruh University
Locations (1):
- Artvin State Hospital, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kizkin ZY, Oguz S, Ak S. The Effect of Graded Motor Imagery on Pain and Function in Individuals With Knee Osteoarthritis: A Comparative Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Jun 1;104(6):534-543. doi: 10.1097/PHM.0000000000002663. Epub 2024 Nov 28. PMID 39642317

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05925517/Prot_SAP_000.pdf